CLINICAL TRIAL: NCT01227434
Title: A Phase II Study of PD 0332991 in Patients With Recurrent Rb Positive Glioblastoma
Brief Title: A Study of PD 0332991 in Patients With Recurrent Rb Positive Glioblastoma
Acronym: PD0332991
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10105
Record Dates: First submitted 2010-10-15; First posted 2010-10-25 (Estimated); Results first posted 2015-06-12 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-06

CONDITIONS: Glioblastoma; Gliosarcoma; Anaplastic Astrocytoma
Keywords: Glioblastoma; Gliosarcoma; Anaplastic astrocytoma; Malignant astrocytoma NOS; Malignant glioma; GBM
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Astrocytoma; Glioma | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical Group (Experimental): PD 0332991 125 mg daily for 7 days prior to an indicated, intended surgical resection as clinical care for progression, and then resume drug at the same dose after recovery from surgery on a repeating schedule of 21 consecutive days of drug followed by a 7 day break off therapy (cycle length is 28 days). Treatment will be repeated every 28 days, and in the absence of disease progression patients may receive treatment for 12 cycles. At that time patients will be given the option to continue on study past 12 cycles, up to a maximum of 24 cycles.
  Interventions: Drug: PD 0332991 (pre-surgery); Drug: PD 0332991; Procedure: Resection as clinical care
- Non-surgical group (Experimental): Patients not in need of surgery treated with PD 0332991 125 mg daily for 21 consecutive days followed by a 7 day break off therapy (cycle length is 28 days). Treatment will be repeated every 28 days, and in the absence of disease progression patients may receive treatment for 12 cycles. At that time patients will be given the option to continue on study past 12 cycles, up to a maximum of 24 cycles.
  Interventions: Drug: PD 0332991

INTERVENTIONS:
Drug: PD 0332991 (pre-surgery) — PD 0332991 for 7 days prior to an indicated, intended surgical resection for progression
  Other Names: Pfizer PD 0332991; palbociclib; IBRANCE, Pfizer, Inc.
  Arms: Surgical Group
Drug: PD 0332991 — PD 0332991 daily for 21 consecutive days followed by a 7 day break off therapy, repeating cycles
  Other Names: Pfizer PD 0332991; palbociclib; IBRANCE, Pfizer, Inc.
Procedure: Resection as clinical care — Indicated, intended, surgical resection as clinical care
  Arms: Surgical Group

SUMMARY:
This study will determine the efficacy of the small molecule CDK4/6 inhibitor PD 0332991 (as measured by progression free survival at 6 months) in patients with recurrent glioblastoma multiforme or gliosarcoma who are Rb positive. A total of 30 patients will be treated; 15 will undergo a planned surgical resection and receive drug for 7 days prior to surgery, followed by drug after recovery from surgery, and the other 15 patients will receive drug without a planned surgical procedure.

DETAILED DESCRIPTION:
A total of 30 patients with recurrent Glioblastoma or Gliosarcoma will be treated with PD 0332991 at a dose of 125 mg daily for 21 consecutive days followed by a 7 day break off therapy (cycle length is 28 days). Of these 30 patients, 15 will receive drug for 7 days prior to an indicated, intended surgical resection for progression, and will then resume drug at the same dose after recovery from surgery. Treatment will be repeated every 28 days, and in the absence of disease progression patients may receive treatment for 12 cycles. At that time patients will be given the option to continue on study past 12 cycles, up to a maximum of 24 cycles.

Following registration, available blocks or slides from a previous surgery must be submitted for diagnosis review (confirmation of Glioblastoma multiforme or Gliosarcoma) and Rb status determination. Only patients with Rb positive tumors can be treated, and Rb tumor status must be known prior to any treatment. Additional tissue from previous surgeries will also be obtained to evaluate molecular abnormalities in the tumor. These studies will be done retrospectively and are not required to be performed prior to registration.

Monitoring will include a clinical and neurological exam before the beginning of each cycle (every 4 weeks). Complete blood counts with differential will be examined on days 1 and 15 of each cycle. Liver and renal function will be performed every 4 weeks. Toxicity and dose modifications will be based on the NCI CTCAE Version 4. Disease status will be assessed clinically each cycle (every 4 weeks) and radiographically after each second cycle (every 8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older with KPS > 60, with life expectancy of > 8 weeks with radiographically proven recurrent, intracranial Glioblastoma multiforme or Gliosarcoma; patients must have documentation of Rb positive disease.
* All patients must sign an informed consent and must have signed an authorization for the release of their protected health information.
* Patients must have had prior external beam radiation and temozolomide chemotherapy; there is no limit to the number of prior chemotherapies used; patients may be treated in their first, second or third relapse
* Patients must have recovered from the toxic effects of prior therapy
* Patients must have adequate bone marrow function and renal function before starting therapy. A pre-study EKG with a normal QT interval is required for all patients
* Patients must have shown unequivocal evidence for tumor progression by MRI scan and on a steroid dose that has been stable for at least 7 days.
* Patients must have an interval of greater than or equal to 42 days from the completion of radiation therapy to study entry.
* A subset of 15 patients will be enrolled prior to a planned, indicated surgical resection. Patients can be enrolled pre-operatively only if they are surgical candidates, do not have evidence of an acute intracranial hemorrhage and are able to start protocol treatment in a window of 7 days before surgery.
* Male and female patients with reproductive potential must use an approved contraceptive method. Women of childbearing potential must have a negative beta-HCG pregnancy test
* Blocks or slides of tumor tissue from a previous surgery must be available to do IHC Rb staining. Patients with negative tumors (Rb negative) will be excluded from the study.

Exclusion Criteria:

* Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
* Patients on enzyme-inducing anti-epileptic drugs or other drugs that cause CYP3A enzyme induction or inhibition will not be eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Prados, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Taylor JW, Parikh M, Phillips JJ, James CD, Molinaro AM, Butowski NA, Clarke JL, Oberheim-Bush NA, Chang SM, Berger MS, Prados M. Phase-2 trial of palbociclib in adult patients with recurrent RB1-positive glioblastoma. J Neurooncol. 2018 Nov;140(2):477-483. doi: 10.1007/s11060-018-2977-3. Epub 2018 Aug 27. PMID 30151703

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 23 participants consented, 1 was found ineligible prior to randomization
Groups:
- Surgical Group: PD 0332991 125 mg daily for 7 days prior to an indicated, surgical resection for progression, and resume drug at the same dose after recovery from surgery on a repeating schedule of 21 consecutive days of drug followed by a 7 day break off therapy (cycle length is 28 days). Treatment repeated every 28 days, and in the absence of disease progression patients may receive treatment for 12 cycles. At that time patients given the option to continue on study past 12 cycles, up to a maximum of 24 cycles.
- Non-surgical Group: Patients not in need of surgery treated with PD 0332991 at a dose of 125 mg daily for 21 consecutive days followed by a 7 day break off therapy (cycle length is 28 days). Treatment repeated every 28 days, and in the absence of disease progression patients may receive treatment for 12 cycles. At that time patients given the option to continue on study past 12 cycles, up to a maximum of 24 cycles.
Period: Overall Study
Arm/Group | Surgical Group | Non-surgical Group
Started | 6 | 16
Completed | 6 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Surgical Group: PD 0332991 125 mg daily for 7 days prior to an indicated, intended surgical resection for progression, and then resume drug at the same dose after recovery from surgery on a repeating schedule of 21 consecutive days of drug followed by a 7 day break off therapy (cycle length is 28 days). Treatment repeated every 28 days, and in the absence of disease progression patients may receive treatment for 12 cycles. At that time patients given the option to continue on study past 12 cycles, up to a maximum of 24 cycles.
- Non-surgical Group: Patients not in need of surgery treated with PD 0332991 125 mg daily for 21 consecutive days followed by a 7 day break off therapy (cycle length is 28 days). Treatment repeated every 28 days, and in the absence of disease progression patients may receive treatment for 12 cycles. At that time patients given the option to continue on study past 12 cycles, up to a maximum of 24 cycles.
- Total: Total of all reporting groups
Arm/Group | Surgical Group | Non-surgical Group | Total
Number analyzed (Participants) | 6 | 16 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 14 | 19
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 3 | 9 | 12
Region of Enrollment [Number; unit: participants]
  United States | 6 | 16 | 22

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Efficacy of the small molecule CDK4/6 inhibitor PD 0332991 in patients with recurrent glioblastoma multiforme or gliosarcoma who are Rb positive was measured by progression free survival. A total of 30 patients was intended to be treated; up to 15 patients were to undergo a planned, intended surgical resection and receive drug for 7 days prior to surgery, followed by drug after recovery from surgery; and up to 15 patients were to receive drug without a planned surgical procedure.
Time Frame: up to 142 weeks
Measure: Mean (Full Range); unit: weeks
Groups:
- Non-surgical Group: Patients not requiring surgery treated with PD 0332991 125 mg daily for 21 consecutive days followed by a 7 day break off therapy (cycle length is 28 days). Treatment repeated every 28 days, and in the absence of disease progression patients may receive treatment for 12 cycles. At that time patients given the option to continue on study past 12 cycles, up to a maximum of 24 cycles.
Arm/Group | Surgical Group | Non-surgical Group
Number analyzed (Participants) | 6 | 16
weeks | 4 [3 to 6] | 14 [1 to 142]
Statistical Analysis 1: Comparison: Surgical Group vs Non-surgical Group; Compared to historical estimates of PFS-6 months. With 30 patients, there would be 90% power to detect an improvement in the PFS-6 months rate from 10% (historical estimate) to 30% based on a one-sided exact test with alpha=0.1; Test type: Superiority or Other; p = 0.10, Exact binomial distribution; Exact binomial distribution = 0.10

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: The number of participants with protocol related toxicity described by CTCAE version 4.0
Time Frame: 1-2 years
Measure: Number; unit: participants
Groups:
- Surgical Group: PD 0332991 at a dose of 125 mg daily for 7 days prior to an indicated, intended surgical resection for progression, and then resume drug at the same dose after recovery from surgery on a repeating schedule of 21 consecutive days of drug followed by a 7 day break off therapy (cycle length is 28 days). Treatment repeated every 28 days, and in the absence of disease progression patients may receive treatment for 12 cycles. At that time patients given the option to continue on study past 12 cycles, up to a maximum of 24 cycles.
Arm/Group | Surgical Group | Non-surgical Group
Number analyzed (Participants) | 6 | 16
participants | 6 | 16

ADVERSE EVENTS:
Time Frame: 3 years
Description: Adverse events were collected from date of first drug, until 30 days following completion of study treatment
Arm/Group | Surgical Group | Non-surgical Group
Serious Adverse Events (participants affected / at risk) | 5/6 | 4/16
Other Adverse Events (participants affected / at risk) | 4/6 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgical Group (N=6) | Non-surgical Group (N=16)
Death NOS (General disorders) | 1 (1) | 2 (2) — Not related to study drug
Meningitis (Infections and infestations) | 1 (1) | 0 (0) — Not related to study drug
Wound Infection (Infections and infestations) | 1 (2) | 0 (0) — Not related to study drug
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Not related to study drug
Cerebral Spinal Fluid Leakage (Nervous system disorders) | 1 (1) | 0 (0) — Not related to study drug
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) — Not related to study drug
Headache (Nervous system disorders) | 2 (2) | 1 (1) — Not related to study drug
Seizure (Nervous system disorders) | 2 (2) | 0 (0) — Not related to study drug
Peripheral Motor Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) — Not related to study drug
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Not related to study drug
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Possibly related
Lung Infection (Infections and infestations) | 0 (0) | 1 (1) — Probably related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Surgical Group (N=6) | Non-surgical Group (N=16)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 2
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Cushingoid (Endocrine disorders) | 0 | 1
Blurred vision (Eye disorders) | 1 | 0
Right upper quadrant defect (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Stool urgency (Gastrointestinal disorders) | 0 | 1
Food craving (Gastrointestinal disorders) | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1
Mucositis Oral (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2
Death NOS (General disorders) | 1 | 2
Edema limbs (General disorders) | 1 | 1
Fatigue (General disorders) | 2 | 7
Flu like symptoms (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 2
Groin pain (General disorders) | 0 | 2
Bronchial infection (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 7
Neutrophil count decreased (Investigations) | 0 | 8
Platelet count decreased (Investigations) | 1 | 5
Weight gain (Investigations) | 0 | 2
White blood cell decreased (Investigations) | 0 | 5
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle weakness-left sided (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 2
Hip and shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in chest and shoulder-from fall (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 2
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 2 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Dysphasia (Nervous system disorders) | 1 | 3
Facial nerve disorder (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 2 | 8
Hydrocephalus (Nervous system disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 3
Trouble reading (Nervous system disorders) | 0 | 1
Neglect (Nervous system disorders) | 0 | 1
Decreased coordination (Nervous system disorders) | 0 | 1
L UQ VF neglect (Nervous system disorders) | 0 | 1
Intraventricular hemorrhage (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 2 | 0
Spasticity (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 3
Confusion (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 3
Urinary frequency (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 3
Urinary urgency (Renal and urinary disorders) | 0 | 1
Painful lump (Reproductive system and breast disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Strial rash (Skin and subcutaneous tissue disorders) | 0 | 1
Minor skin changes (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
Deep vein thrombosis (DVT) (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No